CLINICAL TRIAL: NCT05304312
Title: The Role of Kegel Exercises Book to Improve Treatment in Stress Urinary Incontinence Women by Increasing the Adherence
Brief Title: The Role of Kegel Exercises Book to Improve Treatment in Stress Urinary Incontinence Women
Acronym: ROSEBOOK-SUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Surahman Hakim, Head of Urogynecology Department, Indonesia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-09-1140
Record Dates: First submitted 2022-01-26; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stress Urinary Incontinence
Keywords: Kegel Exercises; Compliance; Stress Urinary Incontinence; Pelvic Floor Muscle Traning; IIQ-7; UDI-6; Adherence; Perineometry
MeSH Terms: conditions — Urinary Incontinence, Stress; Patient Compliance

STUDY DESIGN:
Intervention Model Description: There are two groups in which one group will be given a Kegel Exercises guidebook and another group or control will not be given the book. Both groups were equally followed-up for 3 months and examined by UDI-6, IIQ-7, Perineometer, and 1-hour pad test.
Who Masked: Participant
Masking Description: Participants that received the book (intervention) is followed up with different days and different hospitals with patients that were not receiving any book (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with Kegel Exercises book (Experimental): We gave the patient the Kegel Exercises guidebook for them to study, follow, and keep track of their exercise.
  The Kegel Exercises regiment was 10 each slow and fast-twitch muscle contraction for a session. Three sessions a day needed to be done every day for 12 weeks.
  Interventions: Device: Kegel Exercises guidebook
- Women without Kegel Exercises book (No Intervention): We did not give the Kegel Exercises guidebook for the patients We taught the same Kegel Exercises regiment that was 10 each slow and fast-twitch muscle contraction for a session. Three sessions a day and needed to be done every day for 12 weeks

INTERVENTIONS:
Device: Kegel Exercises guidebook — The Kegel exercises book is consisted of basic explanation about stress urinary incontinence and Kegel exercises, how to do Kegel exercises, table for them to write how many session they did in a day, and lastly their report progress (UDI-6, IIQ-7, periineometer, and 1-hour pad test) that we updated every four weeks
  Arms: Women with Kegel Exercises book

SUMMARY:
This research aims to evaluate a Kegel Exercises guidebook to treat stress urinary incontinence (SUI) in female patients. The Kegel Exercises guidebook had been made and evaluated before, this was a clinical trial to test out the book in clinical settings. In measuring the effectiveness of the book, the investigators used some examinations and questionnaires such as UDI-6, IIQ-7, perineometer, and 1-hour pad test improvement. Investigators followed up the patient's symptoms subjectively with UDI-6 and IIQ-7 and objectively with a perineometer and 1-hour pad test every four weeks.

DETAILED DESCRIPTION:
This research aims to evaluate the Kegel Exercises guidebook in treating stress urinary incontinence in female patients. The guidebook had been produced through rigorous previous research with many evaluations from many clinicians, urogynecologists, and patients. The editing and evaluation process took some time and before long the guidebook was ready to be tested in the clinical setting.

The Investigators enrolled 85 patients in the intervention group and 85 patients in the control group after population sampling calculation. The patients in the intervention group were supervised by the Kegel guidebook however, the patients in the control group were supervised without the Kegel guidebook. The patients in the intervention group were enrolled from Cipto Mangunkusumo Hospital and YPK Mandiri Hospital. For the control group, the investigators enrolled the patients from Buah Hati Hospital and Fatmawati Hospital. Investigators enrolled the patients from different hospitals to mask the book as the intervention to the patients.

The Kegel regiment the Investigators taught were the same. The exercises consisted of two types of movements that contracted the fast-twitch muscle and the slow-twitch muscle. The Investigators recommended doing the fast repetitions ten times a session and the slow repetitions ten times a session. The patients needed to do three sessions for a day, and every day for a week.

To examine the improvement of the symptoms, the investigators used many parameters such as UDI-6 and IIQ-7 questionnaire, a perineometer, and a 1-hour pad test. The investigators evaluate the parameters before the therapy and followed them every four weeks up until 12 weeks of follow-up. The investigators also count how many kegel exercises they did in four weeks, by checking on their Kegel exercises book or by recalling method in control group

ELIGIBILITY:
Inclusion Criteria:

* Women with Stress Urinary Incontinence
* Good cognitive function (based on Moca-Ina questionnaire > 26)
* Able to do Kegel Exercises without restrictions
* Signed the informed consent form

Exclusion Criteria:

* Patient that had incontinence surgery before or other incontinence therapy other than Kegel exercises
* Mix urinary incontinence
* abnormal uterine bleeding
* Pelvic organ prolapse >2 stage
* a severe neurological disorder
* active urinary tract infections
* malignancy on pelvic
* Trauma or radiation therapy on pelvic
* Had other risk factors that may influence persistent high abdominal pressure

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Compliance | up to 12 weeks
  We expect that the patients did a total of 1000 contractions slow and fast twitch muscle. Patients that did less than 1000 contractions a month are classified as non-comply. On the other hand patients who had done 1000 or more contractions were classified as comply
Treatment Success | up to 12 weeks
  Decrease of symptoms based on UDI-6
Treatment Success | up to 12 weeks
  Decrease of symptoms based on IIQ-7
Treatment Success | up to 12 weeks
  Decrease of symptoms based on 1-hour pad test

SECONDARY OUTCOMES:
Improvement of Pelvic floor muscle strength | up to 12 weeks
  measuring the pelvic floor muscle tone at rest and maximum squeeze (min 0) and a higher score means higher muscle tone produced

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Andersson KE, Birder L, Brubaker L, Cardozo L, Chapple C, Cottenden A, Davila W, de Ridder D, Dmochowski R, Drake M, Dubeau C, Fry C, Hanno P, Smith JH, Herschorn S, Hosker G, Kelleher C, Koelbl H, Khoury S, Madoff R, Milsom I, Moore K, Newman D, Nitti V, Norton C, Nygaard I, Payne C, Smith A, Staskin D, Tekgul S, Thuroff J, Tubaro A, Vodusek D, Wein A, Wyndaele JJ; Members of Committees; Fourth International Consultation on Incontinence. Fourth International Consultation on Incontinence Recommendations of the International Scientific Committee: Evaluation and treatment of urinary incontinence, pelvic organ prolapse, and fecal incontinence. Neurourol Urodyn. 2010;29(1):213-40. doi: 10.1002/nau.20870. No abstract available. PMID 20025020
- [Background] Rivas Alonso A, Franquet Casas T, Arellano Atienza P, Berdusan Sanchez M. [Wunderlich disease. First manifestation of a renal adenocarcinoma]. Arch Esp Urol. 1992 Jan-Feb;45(1):73-5. Spanish. PMID 1586224
- [Background] Imamura M, Hudson J, Wallace SA, MacLennan G, Shimonovich M, Omar MI, Javanbakht M, Moloney E, Becker F, Ternent L, Montgomery I, Mackie P, Saraswat L, Monga A, Vale L, Craig D, Brazzelli M. Surgical interventions for women with stress urinary incontinence: systematic review and network meta-analysis of randomised controlled trials. BMJ. 2019 Jun 5;365:l1842. doi: 10.1136/bmj.l1842. PMID 31167796
- [Background] Bo K. Pelvic floor muscle training is effective in treatment of female stress urinary incontinence, but how does it work? Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):76-84. doi: 10.1007/s00192-004-1125-0. Epub 2004 Jan 24. PMID 15014933
- [Background] Borello-France D, Burgio KL, Goode PS, Ye W, Weidner AC, Lukacz ES, Jelovsek JE, Bradley CS, Schaffer J, Hsu Y, Kenton K, Spino C; Pelvic Floor Disorders Network. Adherence to behavioral interventions for stress incontinence: rates, barriers, and predictors. Phys Ther. 2013 Jun;93(6):757-73. doi: 10.2522/ptj.20120072. Epub 2013 Feb 21. PMID 23431210
- [Background] Felicissimo MF, Carneiro MM, Saleme CS, Pinto RZ, da Fonseca AM, da Silva-Filho AL. Intensive supervised versus unsupervised pelvic floor muscle training for the treatment of stress urinary incontinence: a randomized comparative trial. Int Urogynecol J. 2010 Jul;21(7):835-40. doi: 10.1007/s00192-010-1125-1. Epub 2010 Feb 24. PMID 20179901
- [Background] Asklund I, Nystrom E, Sjostrom M, Umefjord G, Stenlund H, Samuelsson E. Mobile app for treatment of stress urinary incontinence: A randomized controlled trial. Neurourol Urodyn. 2017 Jun;36(5):1369-1376. doi: 10.1002/nau.23116. Epub 2016 Sep 9. PMID 27611958